CLINICAL TRIAL: NCT04918407
Title: Effects of Empagliflozin in Reducing Oxidative Stress of Diabetic Recipients After Kidney Transplantation
Brief Title: Effects of Empagliflozin in Reducing Oxidative Stress After Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBMU98543
Record Dates: First submitted 2021-05-29; First posted 2021-06-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — empagliflozin; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Adding 25mg Empagliflozin on Insulin
  Interventions: Drug: Empagliflozin 25 MG; Drug: Insulin
- Insulin alone (Active Comparator): Just contriling the blood glucose with Insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Empagliflozin 25 MG — 25 mg
  Arms: Empagliflozin
Drug: Insulin — Insulin

SUMMARY:
The purpose of this study is to investigate the effect of empagliflozin on oxidative stress in patients with type 2 diabetes after kidney transplantation. The association is examined by comparing the difference in oxidative modifications before and after 90 days treatment with 25 mg empagliflozin plus insulin compared to insulin treatment. The study is randomised and double-blinded. Each treatment group consists of 20 patients. Oxidative stress markers are measured by serum level of superoxide dismutase activity ,lipid peroxidation assay kit, glutathione assay, glutathione peroxidase activity , total antioxidant capacity assay oxidant status , carbonyl content assay and bca protein assay . . A student t-test will be performed to compare adding empagliflozin . The results will be published in a peer-review journal.

DETAILED DESCRIPTION:
With the purpose of studying the antioxidant activity of empagloflozin 25mg will add on insulin in 20 patients after kidney transplant and will compare with 20 diabetic recipient of kidney transplant on insulin therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* HbA1c: 6.5-9.0%
* post kidney transplant
* stable graft function

Exclusion Criteria:

* pancreas and kidney transplant
* history of recurrent urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
serum level of superoxide dismutase | Change from baseline after 90 days of intervention
  Serum level of antioxidant levels

SECONDARY OUTCOMES:
Plasma levels of malondialdehyde | Change from baseline after 90 days of intervention
  Serum level of antioxidant levels

CONTACTS AND LOCATIONS:
Overall Officials: Nooshin Dalili, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (2):
- Iran (2):
  - Labbafinezhd Hospital, Tehran
  - SBMU, Tehran

IPD SHARING:
Plan to Share IPD: No